CLINICAL TRIAL: NCT03978923
Title: Observational Study on the Preparation of the Implant Site With Piezosurgery vs Drill: Comparison Between the Two Methods in Terms of Post-operative Pain, Surgical Times and Operational Advantages
Status: Completed | Type: Observational
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Bevilacqua Lorenzo, prof, University of Trieste
Other Study IDs: UTrieste1
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Preparation of the Implant Site With Piezosurgery vs Drill
Keywords: ultrasonic surgery; piezosurgery; implant bed preparation; microcracks; pain; crestal bone resorption
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the drill-inserted implants (G1)
  Interventions: Device: preparation of the implant site with Piezosurgery vs drill
- the ultrasonic device- inserted implants (G2)
  Interventions: Device: preparation of the implant site with Piezosurgery vs drill

INTERVENTIONS:
Device: preparation of the implant site with Piezosurgery vs drill — The surgery was always performed by the same operator (M.M.) to reduce the bias of the study. Loco-regional anesthesia was performed with Mepivacaine hydrochloride with 1:100000 adrenaline.
  For the preparation of implant sites using traditional methods, the drills were used following manufacturer's protocol by the implant system in use (WINSIX®- BioSAF IN s.r.l, Trezzano Rosa, Trezzano Rosa, Milano - Italy).
  For the preparation of sites was used ultrasonic device, (Surgysonic II, Esacrom S.r.l., Imola, Italy). For the final preparation and insertion of implants, 5-6 ultrasound inserts were used in sequence as follows: tip-shape 1st insert (ES012X) and 2nd insert (ES052XG), crown-shape 3rd insert (ES040), 4th insert (ES041), 5 ° insert (ES043) and 6th insert (ES044).
  The implant insertion was performed with a maximum torque of 35 Ncm. Finally, the cap screws were positioned, and the flaps were sutured in Vycril® 3.0.

SUMMARY:
Purpose: Recent advances showed that ultrasonic implant site osteotomy is related with a decreased trauma and a better post operative healing of the surgical site if compared to the traditional drilling techniques. The micrometric bone cutting control and the operative advantages related to the piezoelectric approach is also characterized by a learning curve for the clinician in surgical practice and an increased operative duration of the procedure. The aim of this investigation was to compare the operative time, the post operative pain and the patients frequency of intake of painkillers in the healing period.

Methods: A total of 75 patients were treated at the Unit of Oral Surgery (Department of Medical Sciences, Surgery and Health, University of Trieste, Italy) in a split mouth model: 75 drill-inserted implants (G1) and 75 piezoelectric device- inserted implants (G2). The Visual Analogue Scale (VAS) was performed to evaluate the post-operative pain at 15 days from the surgery. The operative time and frequency of intake of painkillers was measured.

DETAILED DESCRIPTION:
Materials and Methods The study was conducted after the approval of the local ethical Comettee (n. 88-10.05.2018) University of Trieste.

The following study took into account adult patients undergoing implant therapy with insertion of two contralateral conical implants with a diameter between 3.8 and 4.5 mm with a maximum torque of 35 Ncm. One site was prepared with Ultrasonic device (Esacrom, Imola, Italy) while the contralateral was prepared with micromotor and dedicated drills. All patients were treated at the Unit of Oral Surgery (Department of Medical Sciences, Surgery and Health, University of Trieste, Italy). Seventy-five patients were enrolled in the study, 44 women and 31 men, aged between 45 and 70, who underwent implant therapy in the period between January 2013 and December 2017. The inclusion criteria were: edentulous or partly edentulous with a bilateral loss of teeth in the maxillary or mandible and bone type D2 or D3, following Misch classification16.

The exclusion criteria included: general contraindications to implant surgery, severe coagulation disorders, leukocyte or metabolic diseases, immunosuppressed or immunocompromised patients, patients receiving chemotherapy for less than 1 year, patients on therapy or having taken amino- bisphosphonates intravenously, patients irradiated to the head or neck, patients with uncontrolled diabetes, pregnant and lactating patients, patients with poor oral hygiene and motivation, patients needing maxillary sinus lift concomitant with implant insertion, post-extraction sites with acute or purulent infections.

The final sample of the implants inserted was 150 (75 per technique) then identifying two dependent groups: the drill-inserted implants (G1) and the ultrasonic device- inserted implants (G2). Each patient subscribed an informed written consent and underwent a pre-operative oral hygiene session. Two grams of Amoxicillin were administered to each patient in the preoperative phase. Before surgery, each patient made a rinse with a 0.2% chlorhexidine mouthwash for one minute. The surgery was always performed by the same operator (M.M.) to reduce the bias of the study. Loco-regional anesthesia was performed with Mepivacaine hydrochloride with 1:100000 adrenaline.

For the preparation of implant sites using traditional methods, the drills were used following manufacturer's protocol by the implant system in use (WINSIX®- BioSAF IN s.r.l, Trezzano Rosa, Trezzano Rosa, Milano - Italy).

For the preparation of sites was used ultrasonic device, (Surgysonic II, Esacrom S.r.l., Imola, Italy). For the final preparation and insertion of implants, 5-6 ultrasound inserts were used in sequence as follows: tip-shape 1st insert (ES012X) and 2nd insert (ES052XG), crown-shape 3rd insert (ES040), 4th insert (ES041), 5 ° insert (ES043) and 6th insert (ES044).

The implant insertion was performed with a maximum torque of 35 Ncm. Finally, the cap screws were positioned, and the flaps were sutured in Vycril® 3.0.

Each patient was prescribed a 0.2% chlorhexidine mouthwash to be used twice a day for two weeks and paracetamol 1000 mg (maximum 3 tablets a day) as a pain-relieving therapy.

Each patient included in the study was therefore in possession of two questionnaires, one per technique, for the evaluation of the treatment. In the questionnaire the patient was asked to trace an "X" representing the level of pain experienced. The questionnaire recorded the individual symptoms experienced during the surgery, after 8 hours, from the 1st to the 7th day and finally any persistence

of the symptoms on the 15th day after surgery. In the same questionnaire was also asked to indicate the possible intake of painkillers and the related dose, after surgery and in the following six days; moreover, after the fifteenth day, the patient was asked if he have repeated the experience of the implant surgery. Then, for each patient, a postoperative check was scheduled: after one week all the patients were recalled for a post-operative control and the removal of the sutures.

For the subjective analysis of the effects of the two methods, it was decided to use the Visual Analogue Scale (VAS). This linear scale is the visual representation of the amplitude of pain that the patient perceives. It is a horizontal line 100 mm long, in which one end indicates the absence of pain, while the other represents the worst pain imaginable.

During the surgical procedure the preparation times of the implant site were measured from the preparation of the flap up to the insertion of the implant.

Immediately after the end of the surgical procedure, a questionnaire on the operative difficulty was compiled by the operator. In particular, the two techniques were compared considering two factors: the easiness in obtaining a correct axis of implants insertion and the quality of visibility. Furthermore, a cumulative judgement has been done for the whole procedure, as "simple", "of medium difficulty", "difficult".

Statistical Analysis SPSS software (SPSS Inc. Chicago, IL) was used for statistical analysis. A value of p <0.05 was used in rejecting the null hypothesis.

In addition, continuous data were analyzed using non-parametric tests given the asymmetric distribution of some data sets.

Friedman test was used to evaluate the significance of VAS differences within groups over time. Wilcoxon test was used to evaluate the significance of VAS differences within groups and between groups at each time point.

A Cochrane test was used to assess the significance of differences in the frequency of intake of painkillers within groups over time. Subsequently, a McNemar test was used for post-hoc analysis and to assess the significance of differences in the frequency of intake of painkillers between groups each time point.

After having calculated the mean operative times for G1 and G2 Mann-Whitney test was used to compare the differences in surgical times between D2 and D3 bone type within each group while Wilcoxon test was used to intercept the differences between groups in bone type D2 and D3, respectively.

The same McNemar test was used to test the differences in the operator questionnaire answers between groups.

ELIGIBILITY:
Inclusion Criteria:

* edentulous or partly edentulous with a bilateral loss of teeth in the maxillary or mandible
* bone type D2 or D3, following Misch classification

Exclusion Criteria:

* general contraindications to implant surgery
* severe coagulation disorders
* immunosuppressed or immunocompromised patients
* patients receiving chemotherapy for less than 1 year
* patients on therapy or having taken amino-bisphosphonates intravenously
* patients irradiated to the head or neck
* patients with uncontrolled diabetes
* pregnant and lactating patients
* patients with poor oral hygiene and motivation
* patients needing maxillary sinus lift concomitant with implant insertion
* post-extraction sites with acute or purulent infections.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: . Seventy-five patients were enrolled in the study, 44 women and 31 men, aged between 45 and 70
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
level of pain experienced | 1.1.2013-31.12.2017

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Sciences, University of Trieste, Trieste, Italy, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maglione M, Bevilacqua L, Dotto F, Costantinides F, Lorusso F, Scarano A. Observational Study on the Preparation of the Implant Site with Piezosurgery vs. Drill: Comparison between the Two Methods in terms of Postoperative Pain, Surgical Times, and Operational Advantages. Biomed Res Int. 2019 Sep 29;2019:8483658. doi: 10.1155/2019/8483658. eCollection 2019. PMID 31662998